CLINICAL TRIAL: NCT00862264
Title: A 12-week Phase III Study to Evaluate the Efficacy and Tolerability of Beclomethasone Dipropionate/Formoterol Single Inhaler HFA 134a-pMDI in Adult Patients With Mild to Moderate Persistent Asthma
Brief Title: Efficacy and Tolerability of Beclomethasone Dipropionate/Formoterol Single Inhaler in Patients With Mild to Moderate Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA/PR/033011/005/04; 2004-000718-37 (EudraCT Number)
Record Dates: First submitted 2009-02-25; First posted 2009-03-16 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF 1535 pMDI (Experimental): CHF 1535 HFA pMDI aerosol (100 µg/unit dose of beclomethasone dipropionate plus 6 µg of formoterol/unit dose
  Interventions: Drug: Fixed combination Beclomethasone Dipropionate/Formoterol HFA 134a-pMDI
- BDP pMDI (Active Comparator): Beclomethasone dipropionate-CFC pMDI, 250 µg/unit dose
  Interventions: Drug: Fixed combination Beclomethasone Dipropionate/Formoterol HFA 134a-pMDI

INTERVENTIONS:
Drug: Fixed combination Beclomethasone Dipropionate/Formoterol HFA 134a-pMDI — Fixed combination Beclomethasone Dipropionate/Formoterol HFA 134a-pMDI

SUMMARY:
Efficacy and tolerability of the fixed combination Beclomethasone Dipropionate /Formoterol in patients with mild to moderate persistent asthma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and tolerability of Beclomethasone Dipropionate/Formoterol single inhaler in a twice daily regimen in patients with mild to moderate persistent asthma. Patients are randomised to receive either Beclomethasone Dipropionate/ formoterol single inhaler (total daily dose : BDP/FF 400/24 µg) or Beclomethasone CFC (total daily dose : BDP 1000 µg) during 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate persistent asthma (according to GINA 2003 guidelines)
* FEV1 > or = 60% and < or = 85% of predicted normal values
* Patients free of LABA at least for one month before screening and already treated for at least two months with ICS and experiencing (i)a daily use of SABAs between 1 and 4 puffs, (ii) and/or clinical symptoms three times in the week prior to inclusion
* A documented positive response to the reversibility test

Exclusion Criteria:

* Pregnant or lactating females or women of childbearing potential without any efficient contraception
* Heavy smokers defined as smoking for > 10 pack years
* Evidence of asthma exacerbation causing an hospitalisation or requiring treatment with oral/parenteral corticosteroids or evidence of symptomatic airways infection in the 4 weeks prior to inclusion (3 months for slow-release corticosteroids)
* Seasonal asthma or asthma occurring only during episodic exposure to an allergen or occupational chemical sensitizer
* Clinical significant or unstable concomitant diseases, including clinically significant laboratory abnormalities
* Evidence of asthma worsening during the week preceding randomisation (e.g PEF variability > or = 30% during 2 consecutive days, SABA use > 8 puffs/day during 2 consecutive days, nocturnal awakenings due to asthma symptoms during 3 consecutive days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2004-08; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Pre-dose morning PEF | At the end of treatment after 3 month of treatment

SECONDARY OUTCOMES:
Pre-dose FEV1 - Other spirometric parameters - | Every 6 weeks
Percentage of night and/or days free of clinical symptoms | End of treatment after 3 month of treatment
Morning and evening asthma clinical symptom scores | End of treatment after 3 month of treatment
Use of rescue short-acting b2-agonists | End of treatment after 3 month of treatment
Asthma exacerbations | Every 6 weeks
Safety and Tolerability | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Bonnet Gonod, Study Director — Chiesi Farmaceutici

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2004-000718-37